CLINICAL TRIAL: NCT03431064
Title: Lung Recruitment Maneuver as a Potential Predictor of Fluid Responsiveness in Mechanically Ventilated Pediatric Patients
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Masimo Corporation (Industry)
Responsible Party: Principal Investigator, Viviane Nasr, Cardiac Anesthesiologist, Boston Children's Hospital
Other Study IDs: IRB-P00025702
Record Dates: First submitted 2018-02-02; First posted 2018-02-13 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Anesthesia; Intravenous Fluid; Blood Pressure
MeSH Terms: interventions — Hypodermoclysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical patients less than 18 years old: Patients less than 18 years old having surgery with general anesthesia at Boston Children's Hospital
  Interventions: Other: Lung Recruitment Maneuver; Other: Fluid Administration

INTERVENTIONS:
Other: Lung Recruitment Maneuver — Lung Recruitment Maneuver by Anesthesiologist
Other: Fluid Administration — Administration of IV Fluid by Anesthesiologist

SUMMARY:
In this research study we want to learn more about using non-invasive tools as a way to predict whether or not a child under general anesthesia will require and respond to fluid administration.

It is important for an anesthesiologist to know if a child would respond to fluid administration so that they can provide the optimal intervention for low blood pressure and avoid unnecessary treatment.

DETAILED DESCRIPTION:
In this research study we want to learn more about using non-invasive tools as a way to predict whether or not a child under general anesthesia will require and respond to fluid administration.

It is important for an anesthesiologist to know if a child would respond to fluid administration so that they can provide the optimal intervention for low blood pressure and avoid unnecessary treatment.

ELIGIBILITY:
Inclusion Criteria:

* 0 to < 18 years old
* Undergoing surgery at Boston Children's Hospital under general anesthesia
* mechanically ventilated with an endotracheal tube
* Monitored with an indwelling radial arterial catheter as part of the anesthetic plan for the scheduled surgical procedure

Exclusion Criteria:

* Prematurity
* Low birth weight
* Congenital heart disease
* Left or right ventricular dysfunction
* Cardiac arrhythmia
* Pulmonary hypertension
* Preoperative parenchymal or interstitial lung disease
* Intracranial hypertension
* Poor transthoracic acoustic window
* Obesity
* Allergy to ultrasound transmission gel
* Need for single lung ventilation
* Systemic hypertension on antihypertensive medications

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Patients less than 18 years old who are scheduled to undergo surgery with general anesthesia at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2018-06-21 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in stroke volume | immediately before and after each intervention
  Evaluate Lung Recruitment Maneuver as a means to predict fluid responsiveness in mechanically ventilated pediatric patients in the operating room.

SECONDARY OUTCOMES:
Change in arterial compliance effect on Systolic Pressure Variation (mmHg) | immediately before and after each intervention
  Evaluate the effect of arterial stiffness on Systolic Pressure Variation (mmHg) in mechanically ventilated pediatric patients in the operating room.
Change in arterial compliance effect on Pulse Pressure Variation (%) | immediately before and after each intervention
  Evaluate the effect of arterial stiffness on Pulse Pressure Variation (%) in mechanically ventilated pediatric patients in the operating room.
Change in arterial compliance effect on Plethysmographic Variability Index (%) | immediately before and after each intervention
  Evaluate the effect of arterial stiffness on Plethysmographic Variability Index (%) in mechanically ventilated pediatric patients in the operating room.

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Nasr, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States